CLINICAL TRIAL: NCT02549144
Title: Effects of a Large Increase in Dietary Fats and Cholesterol on HDL Composition and Function in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Professor Andrea Natali, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HDL-DIET
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Lipids
Keywords: HDL biochemical composition and function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat/cholesterol diet (Experimental): High-fat/high-cholesterol (HFHC) normocaloric diet for 14 days.
  Interventions: Dietary Supplement: High fat/cholesterol diet
- Low fat/cholesterol diet (Experimental): Low-fat/low-cholesterol (LFLC) normocaloric diet for 14 days.
  Interventions: Dietary Supplement: Low fat/cholesterol diet

INTERVENTIONS:
Dietary Supplement: Low fat/cholesterol diet — The low fat/cholesterol diet had 10% calories from fat and 150-200 mg of cholesterol per day.
  Arms: Low fat/cholesterol diet
Dietary Supplement: High fat/cholesterol diet — The high fat/cholesterol diet had 40% calories from fat and 250-300 mg of cholesterol per day
  Arms: High fat/cholesterol diet

SUMMARY:
In this study the investigators aimed at measuring the effect of a two-week high-fat/high-cholesterol (HFHC) normocaloric diet on HDL particles biochemical composition and HDL function compared to a two-week low-fat/low-cholesterol (LFLC) normocaloric diet.

DETAILED DESCRIPTION:
HDL particles can change their composition and function in response to a variety of pathological conditions and environmental stimuli. It has been previously shown that a western diet is able to drastically modify biochemical composition, anti-inflammatory and anti-oxidant properties of HDL in animals. In humans little is known on the role of diet on HDL function and composition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 and ≤40 years of age
* Lean or overweight (BMI: 18 to 29,9 kg/m2)
* Normal liver and kidney function
* Normal thyroid function
* Stable weight in the last 3 months
* Read and understood the informed consent form and signed it voluntarily

Exclusion Criteria:

* Liver, heart, kidney, lung, infectious, neurological, psychiatric, endocrine, immunological or neoplastic diseases
* Chronic use of drugs or vitamin supplements
* Smoking
* Pregnancy or lactation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Dichlorofluorescein fluorescence slope | 14 days

SECONDARY OUTCOMES:
hydroxyeicosatetraenoic acid | 14 days
hydroxyoctadecadienoic acid | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, Prof, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

REFERENCES:
- [Derived] Morgantini C, Trifiro S, Trico D, Meriwether D, Baldi S, Mengozzi A, Reddy ST, Natali A. A short-term increase in dietary cholesterol and fat intake affects high-density lipoprotein composition in healthy subjects. Nutr Metab Cardiovasc Dis. 2018 Jun;28(6):575-581. doi: 10.1016/j.numecd.2018.03.005. Epub 2018 Mar 19. PMID 29699812
- [Derived] Trico D, Trifiro S, Mengozzi A, Morgantini C, Baldi S, Mari A, Natali A. Reducing Cholesterol and Fat Intake Improves Glucose Tolerance by Enhancing beta Cell Function in Nondiabetic Subjects. J Clin Endocrinol Metab. 2018 Feb 1;103(2):622-631. doi: 10.1210/jc.2017-02089. PMID 29095990